CLINICAL TRIAL: NCT05772871
Title: Compare the Efficacy and Safety of Prednisone Combined With Huaiqihuang Granule Versus Combined With Levamisole for Primary Nephrotic Syndrome in Children: A Prospective, Multi-center, Randomized, Double-blind, Non-inferiority Study
Brief Title: The Efficacy and Safety of Prednisone Combined With Huaiqihuang Granule for Primary Nephrotic Syndrome in Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jianhua Zhou (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jianhua Zhou, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HQH-202205
Record Dates: First submitted 2023-02-24; First posted 2023-03-16 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Nephrotic Syndrome in Children
Keywords: Huaiqihuang granule; Children; Nephrotic syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Prednisone; Levamisole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone, Huaiqihuang granule, and Levamisole placebo (Experimental): In this group, patients will take Prednisone, Huaiqihuang granule, and Levamisole placebo.
  Interventions: Drug: Huaiqihuang granule; Drug: Prednisone; Drug: Levamisole placebo
- Prednisone, Levamisole, and Huaiqihuang granule placebo (Placebo Comparator): In this group, patients will take Prednisone, Levamisole, and Huaiqihuang granule placebo.
  Interventions: Drug: Prednisone; Drug: Levamisole; Drug: Huaiqihuang Granule placebo

INTERVENTIONS:
Drug: Huaiqihuang granule — Huaiqihuang Granule, oral administration, recommended daily dose: for body weight <10 kg, 5g, twice a day; for 10 kg ≤ body weight <20 kg, 10g, twice a day; for 20 kg≤body weight <30 kg, 15g, twice a day; for 30 kg≤body weight <50 kg, 20g, twice a day; for body weight>50 kg, 30g, twice a day. Continuous medication until the end of the study (6 months), second relapse, development as steroid-resistant, lost to follow-up, withdrawal from the study for any reason, or death, whichever occurs first.
  Arms: Prednisone, Huaiqihuang granule, and Levamisole placebo
Drug: Prednisone — Prednisone, oral administration, recommended dose: 2mg/kg/d (maximum 60 mg/d) for 4 weeks followed by 2 mg/kg (maximum 60mg) on alternate days for the other 4 weeks. If patients have relapsed during reducing dosage or withdrawal, the patients will receive Prednisone for 8 weeks again [2mg/kg/d (maximum 60 mg/d) for 4 weeks followed by 2 mg/kg (maximum 60mg) on alternate days for the other 4 weeks]. If a second relapse is observed, patients will receive immunosuppressants and then withdraw from the trial.
Drug: Levamisole placebo — Levamisole placebo, 1.25 mg/kg. once daily. Continuous medication until the end of the study (6 months), second relapse, development as steroid-resistant, lost to follow-up, withdrawal from the study for any reason, or death, whichever occurs first.
  Arms: Prednisone, Huaiqihuang granule, and Levamisole placebo
Drug: Levamisole — Levamisole, 1.25 mg/kg. once daily. Continuous medication until the end of the study (6 months), second relapse, development as steroid-resistant, lost to follow-up, withdrawal from the study for any reason, or death, whichever occurs first.
  Arms: Prednisone, Levamisole, and Huaiqihuang granule placebo
Drug: Huaiqihuang Granule placebo — Huaiqihuang Granule placebo, oral administration, recommended daily dose: for body weight <10 kg, 5g, twice a day; for 10 kg ≤ body weight <20 kg, 10g, twice a day; for 20 kg≤body weight <30 kg, 15g, twice a day; for 30 kg≤body weight <50 kg, 20g, twice a day; for body weight>50 kg, 30g, twice a day. Continuous medication until the end of the study (6 months), second relapse, development as steroid-resistant, lost to follow-up, withdrawal from the study for any reason, or death, whichever occurs first.
  Arms: Prednisone, Levamisole, and Huaiqihuang granule placebo

SUMMARY:
This non-inferiority study aims to compare the efficacy of Prednisone combined with Huaiqihuang Granule against Prednisone combined with Levamisole in the treatment of primary nephrotic syndrome (PNS) in children.

DETAILED DESCRIPTION:
Nephrotic syndrome (NS) is the most frequent glomerular disease in children, with an incidence of 1.15-16.9 per 100,000 children. Children present with the disease at a median age of 2-3 years, and it is twice as common in boys. More than 90% of children who present with NS respond to corticosteroid treatment, and current practice is to treat most patients empirically with prednisone. However, after initial successful treatment, around 80% of children with steroid sensitive NS have disease relapses requiring further courses of prednisone. About 50% of patients develop frequent relapsing or steroid dependent. Further, the long-term use of corticosteroids is associated with numerous side effects, like obesity, diabetes and hypertension.

Traditional Chinese medicine plays a unique role in the enhancement of immune function and kidney function. Huaiqihuang granule is composed of Trametes robiniophila Murr, Fructus Lycii, and Polygonatum sibiricum. It has been used for the treatment of primary nephrotic syndrome (PNS) in China. Previous studies showed Huaiqihuang granule combined with corticosteroids could significantly decrease relapse and infection rates of PNS and were well tolerated by children. This non-inferiority study aims to compare the efficacy of Prednisone combined with Huaiqihuang Granule against Prednisone combined with Levamisole in the treatment of PNS in children.

In this study, about 20 research centers will participate. A total of 402 participants will be divided into two groups (the intervention group and control group) at a ratio of 1:1. The intervention group will receive Prednisone, Huaiqihuang granule and Levamisole placebo, and the control group will receive Prednisone, Levamisole and Huaiqihuang granule placebo. The planned length of patient recruitment enrolment will be 2 years and the total length of visits be 6 months. After enrollment, participants will be followed up until the end of the study (6 months), second relapse, develop as steroid-resistant, lost to follow-up, withdrawal from the study for any reason, or die, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age from 1.5 to 18 years;
* According to the Evidence-based Guideline for Diagnosis and Treatment of Hormone-sensitive, Relapsed/dependent Nephrotic Syndrome in Children (2016), children diagnosed with PNS;
* At enrollment, estimated glomerular filtration rate (eGFR)≥90ml/min/1.73m2；
* At enrollment, serum albumin level below 30g/L, and morning urine protein is 4+ or urinary albumin/creatinine ratio (ACR)≥2.0g/g;
* Volunteered to participate in this study and signed informed consent. For children less than 8 years, legal guardians need to sign the informed consent.

Exclusion Criteria:

* Children who were diagnosed as steroid-resistant NS;
* Patients who received Prednisone, other corticosteroids (like Prednisolone, Methylprednisolone), or immunosuppressants (Tacrolimus, Mycophenolate Mofetil, Cyclosporine A, Rituximab, Cyclophosphamide) within 3 months before enrollment;
* Secondary NS caused by lupus nephritis, hepatitis B associated nephritis, purpura nephritis, and EB virus, cytomegalovirus (CMV), etc;
* With combined diseases of autoimmune disorder or primary immunodeficiency or malignancy;
* With combined diseases of the cardiovascular, liver, hematopoietic system, mental disorders, and other serious diseases;
* With serious infectious diseases (like tuberculosis) in the past or at present;
* With combined diseases of Human immunodeficiency virus (HIV), hepatitis B and /or C virus (HBV, HCV), and other active virus infections;
* History of diabetes;
* Abnormal liver function: alanine aminotransferase and aspartate aminotransferase levels exceed twice the upper limit of the normal range;
* Participation in other ongoing clinical trials;
* Other reasons that the researcher considers unsuitable to participate in this study.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 402 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Maintaining remission rate | Start of randomization until 6-month follow-up
  At the end of the study, the proportion of patients who maintained urine protein negative without relapse (removed the patients who developed steroid resistance at the first 4 weeks of treatment of Prednisone).

SECONDARY OUTCOMES:
Remission time to first relapse | Start of onset of remission after treatment until first relapse, assessed up to 6-month
  Among patients who get remission after treatment, time from the onset of remission to the first relapse
Number of relapses | Start of randomization until 6-month follow-up
  Among patients who get remission after treatment, number of relapse per patient
Relapse rate | Start of randomization until 6-month follow-up
  Among patients who get remission after treatment, proportion of patients with relapse
Incidence of frequently relapse | Start of randomization until 6-month follow-up
  Among patients who get remission after treatment, proportion of patients with more than two times of relapses within 6-month follow-up
Infection rate | Start of medication until 6-month follow-up
  Proportion of patients experiencing infection during the treatment. Infections include respiratory tract infections, urinary tract infections, skin infections, gastrointestinal infections, and others.
Cumulative corticosteroids dosage adjusted by body weight | Start of receiving corticosteroids until 6-month follow-up
  Total amount of per patient per kilogram cumulative corticosteroids dosage
Change in serum creatinine and estimated glomerular filtration rate (eGFR) before and after treatment | Start of randomization until 6-month follow-up
  The level change of serum creatinine, eGFR between baseline and the last testing result during follow-up
Change in serum albumin before and after treatment | Start of randomization until 6-month follow-up
  The level change of serum albumin between baseline and the last testing result during follow-up
Change in urinary albumin/creatinine ratio (ACR) before and after treatment | Start of randomization until 6-month follow-up
  The level change of urinary albumin/creatinine ratio (ACR) between baseline and the last testing result during follow-up
Change in 24h urinary protein (applying to more than 3 years patients) before and after treatment | Start of randomization until 6-month follow-up
  The level change of 24h urinary protein (applying to more than 3 years patients) between baseline and the last testing result during follow-up
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | Start of randomization until 6-month follow-up
Incidence and severity of adverse reactions (ADR), serious adverse reactions (SADR), suspicious and unexpected serious adverse reactions (SUSAR) | Start of randomization until 6-month follow-up

OTHER OUTCOMES:
Change in blood pressure before and after treatment | Start of randomization until 6-month follow-up
  The level change of blood pressure before and after treatment
Change in height before and after treatment | Start of randomization until 6-month follow-up
  The level change of height before and after treatment
Change in body weight before and after treatment | Start of randomization until 6-month follow-up
  The level change of body weight before and after treatment
Change in BMI before and after treatment | Start of randomization until 6-month follow-up
  The level change of BMI before and after treatment
Change in serum cholesterol before and after treatment | Start of randomization until 6-month follow-up
  The level change of serum cholesterol before and after treatment
Change in serum triglycerides before and after treatment | Start of randomization until 6-month follow-up
  The level change of serum triglycerides before and after treatment
Change in serum immunoglobulin before and after treatment | Start of randomization until 6-month follow-up
  The level change of serum immunoglobulin before and after treatment
Change in cortisolv (collecting at 8 am) before and after treatment | Start of randomization until 6-month follow-up
  The level change of cortisolv (collecting at 8 am) before and after treatment
Change in serum 25-hydroxyvitamin D before and after treatment | Start of randomization until 6-month follow-up
  The level change of serum 25-hydroxyvitamin D before and after treatment
Change in T cell subtypes before and after treatment | Start of randomization until 6-month follow-up
  The level change of T cell subtypes before and after treatment
Change in the nephronectin before and after treatment | Start of randomization until 6-month follow-up
  The level change of nephronectin before and after treatment
Change in the caveolin-1 before and after treatment | Start of randomization until 6-month follow-up
  The level change of caveolin-1 before and after treatment
Change in the heparanase before and after treatment | Start of randomization until 6-month follow-up
  The level change of heparanase before and after treatment
The mutation ratio of single nucleotide polymorphism (SNP) in children and their parents at enrollment. | At enrollment until randomization.
  The testing SNP including rs 2285450, rs 2073901, rs 3129888, rs 4979462 and et al.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Zhou, Dr., Principal Investigator — Tongji Hospital
Locations (26):
- China (26):
  - Anhui Children's Hospital, Hefei, Anhui
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Children's Hospital, Fuzhou, Fujian
  - People's Liberation Army Joint Logistics Force No. 900 Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hebei Children's Hospital, Shijiazhuang, Hebei
  - Harbin Children's Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Children's Hospital, Zhengzhou, Henan
  - The First Affliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Children's Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Baiqiu'en First Hospital of Jilin University, Changchun, Jilin
  - Dalian Women and Children's Medical Centre, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - Shanxi Children's Hospital, Taiyuan, Shanxi
  - West China Second Hospital of Sichuan University, Chengde, Sichuan
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Tianjin Children's Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uiger Municipal People's Hospital, Ürümqi, Xinjiang
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Women's and Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No